**Version Date:** 03/07/2022

**Official Title:** Communicating the Health Risks of Sugar-Sweetened Beverages: A Randomized-controlled Experiment of Different Nutrition Labels on Purchased and

Consumption

**Brief Title:** Online Study of the Effects of Sugary Drink Warning Labels on Consumption

Reason for difference in ICF title and Protocol title: Our study involves minor deception (approved by the IRB). We are interested in the effects of sugary drink warning labels on participant shopping behavior, but we do not reveal the true purpose of the study until after participants complete it so that their typical shopping behavior is not influenced by the knowledge of the study's purpose. For this reason, our protocol has a different title than the consent form.

Version – 2.0 

Title of the Research Study: Understanding online shopping behavior

Principal Investigator: Christina A. Roberto; 423 Guardian Drive, Blockley Hall,

Philadelphia, PA 19104; 215-746-7064; <a href="mailto:croberto@pennmedicine.upenn.edu">croberto@pennmedicine.upenn.edu</a> **Emergency Contact:** Christina A. Roberto; 423 Guardian Drive, Blockley Hall, Philadelphia, PA 19104; 215-746-7064; <a href="mailto:croberto@pennmedicine.upenn.edu">croberto@pennmedicine.upenn.edu</a>

You are being invited to participate in a research study. Your participation is voluntary, and you should only participate if you completely understand what the study requires and what the risks of participation are. You should ask the study team any questions you have related to participating before agreeing to join the study. If you have any questions about your rights as a human research participant at any time before, during or after participation, please contact the Institutional Review Board (IRB) at (215) 898-2614 for assistance.

The research study is being conducted to learn about your experience using an online store over the next four weeks. You are being asked to join this study because you are 18 years of age or older, have a child between the ages of 6-11 years old and are the primary grocery shopper for your family. You read and speak English and have regular Internet access.

If you agree to join the study, you will be asked to complete the following research procedures: Complete an initial survey prior to shopping online. Once the survey is complete you will be required to purchase at least two items from the online store every week for four weeks. At the end of four weeks, you will be asked to complete a final survey.

Your participation will last for approximately four weeks. This study poses minimal risks and no direct benefit to you. Potential risks include breach of confidentially which researchers aim to minimize. Your alternative to being in the study is to not participate in the study.

If you do not understand what you are reading, please call the research team. Please ask the researcher to explain anything you do not understand, including any language contained in this form. Keep this form; in it you will find contact information and answers to questions about the study. You may ask to have this form read to you.

Version – 2.0 

### What is the purpose of the study?

The purpose of the study is to learn about your experience using an online snack store over the next four weeks.

### Why was I asked to participate in the study?

You are being asked to join this study because you are 18 years of age or older and are the primary grocery shopper for your family. You read and speak English and have regular Internet access. It is your choice whether or not to participate. If you choose to participate, you may change your mind and leave the study at any time. Refusal to participate or stopping your participation will involve no penalty or loss of benefits to which you are otherwise entitled.

#### How long will I be in the study?

The study will take place over a period of 4 weeks. Each week you will be required to purchase at least two items from the store.

#### Where will the study take place?

The study will take place entirely online. You will participant by shopping in an online store. Any surveys you complete will also be done online.

#### What will I be asked to do?

You will be asked to complete an initial survey. Once the survey is complete, you will be emailed a web-link and password that will direct you to the store. Each week you will have money added to your online store account and must purchase at least two items (a beverage and a snack) from the store in order to be considered an active participant in the study. You will receive \$15 for weeks 1 and 2 and \$17 for weeks 3 and 4 if you successfully participate each week. You will be asked to shop in the store for a total of four weeks. At the end of four weeks, you will be asked to complete a final survey.

#### What are the risks?

This study poses minimal risks. Potential risks include breach of confidentiality. We aim to minimize this risk. Only the researchers involved in this study and those responsible for research oversight will have access to the identifiable information provided.

#### How will I benefit from the study?

There is no direct benefit to you. However, your participation will help us learn about consumers shopping experiences.

#### Will I receive the results of research testing?

Most tests done in research studies are only for research and have no clear meaning for participants. Individual research results will not be shared with you, but we will mail you a summary of the overall aggregated research findings from the study.

#### What other choices do I have?

Your alternative to being in the study is to not be in the study.

Version – 2.0 

### What happens if I do not choose to join the research study?

You may choose to join the study, or you may choose not to join the study. Your participation is voluntary.

There is no penalty if you choose not to join the research study. You will lose no benefits or advantages that are now coming to you or would come to you in the future. If you are currently receiving services and you choose not to volunteer in the research study, your services will continue.

#### When is the study over? Can I leave the study before it ends?

The study is expected to end after all participants have completed their 4-weeks of using the store and all the information has been collected. The study may be stopped without your consent for the following reasons:

- The PI feels it is best for your safety and/or health-you will be informed of the reasons why.
- You have not followed the study instructions.
- The PI, the sponsor or the Institutional Review Board (IRB) at the University of Pennsylvania can stop the study anytime.

You have the right to drop out of the research study at anytime during your participation. There is no penalty or loss of benefits to which you are otherwise entitled if you decide to do so. Withdrawal will not interfere with your future care.

If you no longer wish to be in the research study, please contact Christina Roberto, PhD, at croberto@pennmedicine.upenn.edu

#### How will confidentiality be maintained, and my privacy be protected?

We will do our best to make sure that the personal information obtained during the course of this research study will be kept private. Only the researchers involved in this study and those responsible for research oversight will have access to the information you provide. However, we cannot guarantee total privacy. Your personal information may be given out if required by law. If information from this study is published or presented at scientific meetings, your name and other personal information will not be used. The Institutional Review Board (IRB) at the University of Pennsylvania will have access to your records. We may also share your information related to this study with other parties including thesis committee and/or other federal agencies.

An exception to confidentiality is if you report child or elder abuse or neglect, or if you report suicidal or homicidal ideation or intent to the research team. Any information about child or elder abuse or intent to harm yourself or others will be reported to the authorities, as required by law.

What may happen to my information collected on this study?

Version – 2.0 

Your information will be de-identified. De-identified means that all identifiers have been removed. The information could be stored and shared for future research in this de-identified fashion. The information may be shared with other researchers within Penn, or other research institutions, as well as pharmaceutical, device, or biotechnology companies. It would not be possible for future researchers to identify you as we would not share any identifiable information about you with future researchers. This can be done without again seeking your consent in the future, as permitted by law. The future use of your information only applies to the information collected on this study.

### Will I have to pay for anything?

It will not cost you anything to participate in this research.

### Will I be paid for being in this study?

On your first week of shopping in the online store, you will receive \$15 in your online store account. This money will be used to purchase at least two items (a beverage and a snack) from the store each week. After purchasing at least two items during the first week, the amount of money in your account will increase by \$15 the following week as an incentive to remain in the study. For each week that you stay in the study and buy at least one snack and one beverage, the money in your account will increase. The amount you receive will increase to \$17 during the third and fourth weeks if you successfully shop each week. At the end of the study, we will ask you to complete a final survey. If you complete this survey, an additional \$20 will be added to your card for completing the study. Any money you do not spend in the online store will be yours to keep at the end of the study.

## Who can I call with questions, complaints or if I am concerned about my rights as a research subject?

If you have questions, concerns or complaints regarding your participation in this research study or if you have any questions about your rights as a research subject, you should speak with the Principal Investigator, Christina Roberto, listed on page one of this form. If a member of the research team cannot be reached or you want to talk to someone other than those working on the study, you may contact the IRB at (215) 898 2614.

If you have any questions or there is something you do not understand, please ask. You will receive a copy of this consent document.

Version – 2.0 